CLINICAL TRIAL: NCT03090620
Title: A Randomized Trial Comparing Physostigmine vs Lorazepam for Treatment of Adolescent Antimuscarinic (Anticholinergic) Toxidrome
Brief Title: Treatment of Adolescent Antimuscarinic (Anticholinergic) Toxidrome
Acronym: TAAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Academy of Clinical Toxicology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-1730
Record Dates: First submitted 2017-03-10; First posted 2017-03-27 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Anticholinergics Toxicity
MeSH Terms: interventions — Physostigmine; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physostigmine (Experimental): Physostigmine 0.02 mg/kg IV bolus (max of 2 mg), which can be repeated at 10 minutes, followed by a 0.02 mg/kg/hr (max of 2 mg/hr) infusion for 4 hours.
  Interventions: Drug: Physostigmine
- Lorazepam (Experimental): Lorazepam 0.05 mg/kg IV bolus (max 2 mg), which can be repeated at 10 minutes if inadequate patient response, followed by a Normal Saline infusion for 4 hours.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Physostigmine — Administration of physostigmine bolus followed by an infusion
  Arms: Physostigmine
Drug: Lorazepam — Administration of lorazepam bolus followed by normal saline infusion
  Arms: Lorazepam

SUMMARY:
Overdose of xenobiotics (antihistamines, antipsychotics, or Jimson Weed) with resulting antimuscarinic toxidrome is a common scenario in medical toxicology. The result of antagonism of muscarinic receptors is a constellation of signs and symptoms (toxidrome): mydriasis, decreased sweat, decreased bowel sounds, agitation, delirium, hallucinations, urinary retention, tachycardia, flushed skin and seizures. Two treatment options are physostigmine or benzodiazepines.

Although the antimuscarinic toxidrome occurs commonly, physostigmine has been used sparingly despite evidence of safety and efficacy. To demonstrate the utility and safety of physostigmine, the investigators propose a randomized clinical trial of physostigmine compared to benzodiazepine for antimuscarinic toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age >=10 and < 18 years
* Present to the Emergency Department or Intensive Care Unit for an antimuscarinic toxidrome from either a pharmaceutical agent such as antihistamine overdose, or natural toxins or products such as Datura stramonium
* Antimuscarinic toxidrome will be defined with at least one central nervous system agitation effect (agitation, delirium, visual hallucinations, mumbling incomprehensible speech), and at least 2 peripheral nervous system adverse effect (mydriasis, dry mucus membranes, dry axillae, tachycardia, decreased bowel sounds).
* Patients will also be required to have a RASS score of +2 to +4 on initial assessment.

Exclusion Criteria:

* History of seizures or seizure during acute clinical course
* History of asthma or wheezing during clinical course Bradycardia (Heart Rate <60)
* Concomitant use of atropine or choline ester or depolarizing neuromuscular blocker during present illness and hospital course
* Diabetes gangrene, known intestinal obstruction or urogenital tract, vagotonic state
* QRS interval > 120 ms on electrocardiogram
* Known to be pregnant at the time of enrollment
* Known ward of the state

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George S Wang, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physostigmine | Lorazepam
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physostigmine | Lorazepam | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (1.4) | 14.4 (1.3) | 13.9 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
Mean Heart Rate [Mean (Standard Deviation); unit: Beats per minute] | 127 (18) | 117 (10) | 122 (14)
Mean Temperature [Mean (Standard Deviation); unit: Celsius] | 37.3 (0.6) | 37.1 (0.5) | 37.2 (0.5)
Mean Respiratory Rate [Mean (Standard Deviation); unit: Respirations per minute] | 29 (7) | 24 (4) | 27 (5)
Mean Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131 (12) | 127 (14) | 129 (13)
Mean Diastolic Blood Pressure [Mean (Standard Deviation); unit: nnHg] | 80 (11) | 88 (17) | 84 (14)
Mean Oxygen Saturations [Mean (Standard Deviation); unit: %Oxygen] | 96 (2) | 97 (3) | 96 (2)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of RASS Score Between Physostigmine and Lorazepam: Before Bolus
Description: Determine the effectiveness of physostigmine as compared with lorazepam for control of antimuscarinic agitation. Richmond Agitation Sedation Scores (RASS) will be compared throughout treatment protocol. The Richmond Agitation-Sedation Scale (RASS) measures sedation and agitation. Possible scores range from -5 (unarousable) to 0 (alert & calm) to +4 (combative). Scores closer to 0 indicate a better outcome for this measurement.
Time Frame: Baseline, immediately before bolus
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physostigmine | Lorazepam
Number analyzed (Participants) | 9 | 10
score on a scale | 1.5 [1 to 2] | 1 [1 to 1.5]

2. Primary Outcome: Comparison of RASS Score Between Physostigmine and Lorazepam: After Bolus
Description: as for outcome 1
Time Frame: Immediately after bolus, up to 10 minutes post-Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physostigmine | Lorazepam
Number analyzed (Participants) | 9 | 10
score on a scale | 0 [0 to 0] | 1 [1 to 2.5]

3. Primary Outcome: Comparison of RASS Score Between Physostigmine and Lorazepam: 4 Hours
Description: as for outcome 1
Time Frame: 4 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physostigmine | Lorazepam
Number analyzed (Participants) | 9 | 10
score on a scale | 0 [0 to 0] | 0.25 [-1.5 to 1.5]

4. Primary Outcome: Comparison of the Effectiveness in Control of Delirium Between Physostigmine and Lorazepam: Before Bolus
Description: Determine the effectiveness of physostigmine as compared with lorazepam in the reversal of antimuscarinic delirium. Confusion Assessment Method for the ICU (CAM-ICU) scores will be evaluated throughout the study. This measurement is a dichotomous outcome ("yes" or "no" for presence of delirium is indicated rather than a score). The number of participants exhibiting delirium is reported.
Time Frame: Baseline, immediately before bolus
Measure: Count of Participants; unit: Participants
Arm/Group | Physostigmine | Lorazepam
Number analyzed (Participants) | 9 | 10
Participants | 9 | 9

5. Secondary Outcome: Safety and Effectiveness of Physostigmine Infusion in the Setting of Antimuscarinic Toxidrome.
Description: Evaluation of clinical antimuscarinic symptoms, along with presence of any adverse effects, during the infusion to report tolerability, safety profile, and effectiveness of the infusion. the number of participants exhibiting adverse events will be reported, by type.
Time Frame: Up to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Physostigmine | Lorazepam
Number analyzed (Participants) | 9 | 10
Participants
  Seizures | 0 | 0
  Bradycardia | 0 | 0
  Bronchorrhea | 0 | 0
  Bronchospasm | 0 | 0
  Diaphoresis | 0 | 0
  Intubation | 0 | 0
  Vomiting | 1 | 1
  Oversedation | 1 | 1

6. Primary Outcome: Comparison of the Effectiveness in Control of Delirium Between Physostigmine and Lorazepam: After Bolus
Description: as for outcome 4
Time Frame: Immediately after bolus, up to 10 minutes post-Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Physostigmine | Lorazepam
Number analyzed (Participants) | 9 | 10
Participants | 4 | 10

7. Primary Outcome: Comparison of the Effectiveness in Control of Delirium Between Physostigmine and Lorazepam: 4 Hours
Description: as for outcome 4
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Physostigmine | Lorazepam
Number analyzed (Participants) | 9 | 10
Participants | 2 | 10

ADVERSE EVENTS:
Time Frame: 4 Hours
Arm/Group | Physostigmine | Lorazepam
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 2/9 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physostigmine (N=9) | Lorazepam (N=10)
Vomitnig (Gastrointestinal disorders) | 1 (1) | 1 (1) — Vomiting during treatment
Oversedation (Nervous system disorders) | 1 (1) | 1 (1) — Sleepiness, oversedation

LIMITATIONS AND CAVEATS:
We had a smaller sample size. All patients in our cohort ingested antihistamines, the majority of which was diphenhydramine. There were no ingestions of other antimuscarinic xenobiotics. Many of the subjects were enrolled during the overnight hours; in addition to the underlying sedation effect of the ingested agent made an assessment of delirium challenging which may have led to more positive delirium scores in both treatment arms. We did not assess efficacy or safety beyond 4 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03090620/Prot_SAP_000.pdf